CLINICAL TRIAL: NCT02509273
Title: A Double Blind, Randomised, Multicentre, Active Controlled, Parallel-group, Phase III Trial to Evaluate the Efficacy, Safety and Pharmacokinetics of Intravenous Clonidine (Hydrochloride) Compared to Midazolam for Sedation in Children From Birth to Less Than 18 Years of Age
Brief Title: Efficacy, Safety and Pharmacokinetic Study of Intravenous Clonidine Versus Midazolam for Sedation in Paediatric Patients
Acronym: CloSed1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Erasmus Medical Center (Other); University of Tartu (Other); Therakind Ltd (Unknown); Gianni Benzi Pharmacological Research Foundation (Other); University College, London (Other); Karolinska Institutet (Other); Univerzita Karlova v Praze (Other); Vereniging Samenwerkende Ouder- En Patientenorganisaties (Unknown); Bambino Gesù Hospital and Research Institute (Other); European Commission (Other); ARNAS Civico Di Cristina Benfratelli Hospital (Other); Servicio Madrileño de Salud, Madrid, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLON01; 2014-003582-24 (EudraCT Number)
Record Dates: First submitted 2015-04-27; First posted 2015-07-28 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Sedation in Intensive Care
MeSH Terms: interventions — Clonidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLONIDINE HYDROCHLORIDE (Experimental): solution for i.v. infusion (maximum 55 μg/kg per day; maximum 7 day treatment)
  Interventions: Drug: Clonidine
- MIDAZOLAM (Active Comparator): solution for i.v. infusion (maximum 5.5 mg/kg per day; maximum 7 day treatment)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Clonidine
  Arms: CLONIDINE HYDROCHLORIDE
Drug: Midazolam
  Arms: MIDAZOLAM

SUMMARY:
Closed1 aims to compare the efficacy, safety and pharmacokinetics of clonidine (hydrochloride) to midazolam in the sedation of ventilated children and adolescents (0-18 years) admitted to a paediatric intensive care unit (PICU) and requiring mechanical ventilation and sedation for at least 24 hours.

In particular, the proportion of subjects with sedation failure at the maximum possible dose (defined within the study protocol) will be measured. Additionally, the safety and tolerability (including withdrawal effects) of clonidine compared to midazolam will be evaluated. A pharmacokinetic-pharmacodynamic relationship of clonidine for sedation in PICU will be established. Genetic polymorphisms of clinical relevance affecting pharmacokinetics, pharmacodynamics and metabolism will be also identified.

Ad hoc paediatric parenteral formulations of clonidine hydrochloride and midazolam will be manufactured. At least 300 subjects will be enrolled from study centres in five European member countries (Czech Republic, Germany, Italy, the Netherlands, and Sweden).

The clinical study will enrol critically ill paediatric patients who require mechanical ventilation and sedation.

Subjects will be closely followed using standard PICU monitoring of vital functions (continuous assessment of heart rate and peripheral arterial oxygen saturation, intermittent assessment of systolic and diastolic blood pressure), intermittent assessment of pain and depth of sedation, documentation of parameters of mechanical ventilation and intermittent arterial blood gas analysis.

The study will be conducted in compliance with the study protocol, Good Clinical Practice (ICH-GCP) and the applicable regulatory requirement(s). In addition, qualified PICU staff will be monitoring subjects around the clock, thus minimising reaction time in case of alarms or deterioration of clinical parameters.

This project has received funding from the European Union's Seventh Framework Programme for research, technological development and demonstration under grant agreement n° 602453.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged from birth (≥34 weeks gestational age [GA]) to <17 years, 11 months, 1 week old
* Admitted or expected to be admitted (post-operatively) to PICU
* Existing or expected indication for invasive or non-invasive ventilation (except Continuous Positive Airway Pressure, CPAP)
* Anticipated need for continuous sedation for at least 24 hours
* Informed consent (or deferred consent) obtained from the subject's parent(s) or legal guardian(s)
* Where applicable, assent obtained from the subject to participate in the clinical trial

Exclusion Criteria:

* Body weight less than 1500 g
* Gestational age [GA] of <34 weeks
* Body weight 3 kg or less AND aged 28 days or older
* Body weight less than 10 kg AND aged 2 years old or older
* Body weight greater than 85 kg
* Subjects who will be 18 years old in less than 3 weeks
* Known hypersensitivity to the IMP (clonidine) or comparator (midazolam), or Non Investigational Medicinal Product (morphine, propofol) or any of their formulation ingredients and their rescue medication
* Subjects anticipated to be treated with forbidden concomitant medications during IMP administration
* Subjects less than 24 hours post-resuscitation
* Subjects who have been under sedation for more than 72 hours immediately prior to assessment
* Subjects currently being treated with Extra Corporeal Membrane Oxygenation (ECMO)
* Subjects with treatment-induced whole body hypothermia
* Subjects with severe organ insufficiencies
* Subjects whose condition is assessed by the investigator to have an effect on the level of consciousness which impairs the assessment of sedation (COMFORT-B/NISS)
* Subjects with phaeochromocytoma
* Subjects with severe bradyarrhythmia resulting from either sick-sinus syndrome or atrioventricular (AV) block of 2nd or 3rd degree
* Known arterial hypertension requiring chronic treatment in medical history
* Females who are pregnant, lactating or planning to become pregnant or who return a positive result to a urine pregnancy test (a dipstick and serum pregnancy test will be performed at the screening visit).
* Employee or direct relative of an employee or any member of the study site staff or the Sponsor/ study management staff (applies to subject and/ or subject's parent(s)
* Participation in a clinical intervention study using drugs within the last 3 weeks
* Previous participation in this clinical study at any time
* Parent(s)/ legal guardian(s) decline to give informed consent. If parent(s)/ legal guardian(s) are not present

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Sedation failure | ≤ 7 days
  measured by pain score Numerical Rating Scale (NRS), sedation score COMFORT-B and sedation score Nurse's Interpretation of Sedation (NISS)

SECONDARY OUTCOMES:
Pharmacokinetics/Pharmacodynamics (PKPD) modeling (measured by plasma concentrations and sedation score results (COMFORT-B) | ≤ 7 days treatment period
  measured by plasma concentrations and sedation score results (COMFORT-B)
Safety assessment (number of patients with adverse events) | ≤ 21 ± 2 days (treatment period, completion visit, post dose monitoring and follow-up visit) in all subjects
  measured by number of patients with adverse events
Extent of withdrawal effects | post dose ≥ 1 day, ≤ 5 days
  measured by score Sophia Observation Withdrawal Symptoms-Paediatric Delirium (SOS-PD)
Extent of rebound hypertension | post dose ≥ 3 days, ≤ 5 days
  measured by blood pressure assessment for at least 72 hours after IMP cessation
Percentage of respiratory depression per group | during re-intubation apnoea in treatment period (≤ 7 days), post dose monitoring every 24 hours up to 10 days
  Number of reintubations / number extubation failures ratio %
Neurodevelopment (Bayley Scales of Infant Development, Second Edition (Bayley-II) score) | 1 year (in neonates only)
  Bayley Scales of Infant Development, Second Edition (Bayley-II) score
Pharmacogenomic assessment (measured by plasma concentrations and candidate gene polymorphisms/genotyping) | On 1 day of treatment period (≤7 days) only
  measured by plasma concentrations and candidate gene polymorphisms/genotyping

CONTACTS AND LOCATIONS:
Locations (10):
- Univerzita Karlova v Praze, Prague, Czechia
- Tallinn Children's Hospital, Tallinn, Estonia
- Germany (2):
  - University of Erlangen-Nürnberg Medical School, Erlangen
  - Diakonie Neuendettelsau - Cnopf'sche Kinderklinik Nürnberg, Nuremberg
- Italy (3):
  - Azienda Ospedaliero Universitaria Policlinico di Bari, Bari
  - ARNAS Civico Di Cristina Benfratelli, Palermo
  - Bambino Gesù Hospital and Research Institute, Rome
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Neubert A, Baarslag MA, Dijk MV, Rosmalen JV, Standing JF, Sheng Y, Rascher W, Roberts D, Winslade J, Rawcliffe L, Hanning SM, Metsvaht T, Giannuzzi V, Larsson P, Pokorna P, Simonetti A, Tibboel D; CLOSED Consortium. The CLOSED trial; CLOnidine compared with midazolam for SEDation of paediatric patients in the intensive care unit: study protocol for a multicentre randomised controlled trial. BMJ Open. 2017 Jun 21;7(6):e016031. doi: 10.1136/bmjopen-2017-016031. PMID 28637741